CLINICAL TRIAL: NCT03909061
Title: Effectiveness of a Remote Wheelchair Maintenance Training Program
Brief Title: Wheelchair Maintenance Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lynn Worobey, Research Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY18100047; 90SI5014-01-00 (Other Grant/Funding Number: Natl Inst on Disability Independent Living and Rehab)
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Remote Maintenance Training Program
Keywords: Wheelchair; Participation; Training; Maintenance; Breakdown
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This is a randomized single blind study.
Masking Description: Subjects will be choose to be in one of three groups: one group will receive maintenance training immediately with no follow up, one group will receive the maintenance training immediate with a 1 month & 6 month follow up, and one group that will be randomized to either receive the maintenance training immediately or to receive the maintenance training after a 6 month wait (with follow ups).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immediate Training (no follow up) (Experimental): Individuals may decide to participate in the research study training program, but not in any follow up questionnaires. This group will have immediate access to the independent maintenance training materials. They will complete data collection measures embedded in the maintenance training program, including demographics, Online Learning Readiness Scale (OLRS), Moorong Self Efficacy Scale (MSES), Patient Reported Outcome Measurement Information System (PROMIS), Assistive Technology Module Questionnaire (ATM-Q), and the Wheelchair Maintenance Training Questionnaire (WMT-Q).
  Interventions: Behavioral: Wheelchair Maintenance Training
- Immediate Training (with follow up) (Experimental): Individuals may decide to participate in the research study, but do not want to be randomized. After consent is obtained, these individuals will be directed immediately to the baseline questionnaires (see above) before and after the wheelchair maintenance training. Participants may also be asked to complete a user satisfaction survey.
  Interventions: Behavioral: Wheelchair Maintenance Training
- Randomized Training (Experimental): Individuals may decide to participate in the research study and agree to be randomized. These individuals will be immediately randomized into an immediate or a wait list control group. The immediate will receive the wheelchair maintenance training program after completing the baseline questionnaires. The wait list control group will wait approximately 6 months before receiving the independent maintenance training program.
  Interventions: Behavioral: Wheelchair Maintenance Training

INTERVENTIONS:
Behavioral: Wheelchair Maintenance Training — Wheelchair Maintenance Training Program: WMTP training consists of three parts. It starts with an overview of basic wheelchair maintenance items, continues with the second section discussing how to inspect the parts of a wheelchair and finishes with the third section discussing how to perform wheelchair maintenance on a wheelchair. Throughout the course, there are videos and pictures demonstrating the activities discussed in the training program. Participants will also be informed when a repair requires professional assistance and where such assistance may be found.

SUMMARY:
The objective of this research study is to assess the effectiveness of a remote wheelchair maintenance training program, and to determine methods which may increase overall success of an online training program.

DETAILED DESCRIPTION:
Up to 100 individuals will be recruited for this research study. We will recruit individuals who use a wheelchair for the majority of their mobility (over 40 hours per week), and have a traumatic spinal cord injury (SCI). This study will be accessed entirely online and participation is expected to last approximately one year. Subjects will select to participate in one of three groups; one group that will receive maintenance training immediately with no follow up, one group that will receive the maintenance training immediately with 1 month and 6 month follow up, and one group that will be randomized to either receive the maintenance training immediately or after 6 months. The maintenance training program itself will take approximately 1-2 hours to complete.

After obtaining informed consent, participants in the first two groups will complete baseline questionnaires. They will then receive the maintenance training program.

Participants in the third group (a wait-list control group) will complete the baseline questionnaires and be contacted one month later to complete a wheelchair maintenance assessment questionnaire. They will then wait 5 months. After this period, participants will complete the baseline questionnaires a second time, and then receive the wheelchair maintenance training.

After completing the maintenance training, all groups will be contacted immediately post training to complete additional questionnaires to assess the effectiveness of the remote training program. Participants in the 2nd and 3rd group will be contacted 1 month and 6 months post-training to complete additional questionnaires. Participants may be compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

* Have a traumatic spinal cord injury
* Use a wheelchair as a primary means of mobility (>40 hours per week)

Exclusion Criteria:

* English is not a primary language
* Primary residence is not in the United States

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Wheelchair Maintenance Training Questionnaire (WMT-Q) | This measure is collected at baseline, pre- training, during the training, as well as at the 1 month and 6 month follow ups.
  The WMT-Q has three sub scales which measure of an individual's knowledge of maintenance (knowledge), their or their caregiver's ability to complete maintenance (capacity), and the frequency at which they or their caregiver perform it (performance). Each subscale ranges from 0-100 with larger numbers indicating greater proficiency.

SECONDARY OUTCOMES:
Change in Assistive Technology Module Questionnaire (ATM-Q) | This measure is collected at baseline, pre- training, and at the 6 month follow up.
  This outcome measure collects information on the number of repairs an individual's wheelchair required as well as the incidence of subsequent consequences from the repair - stranded, injured, missed work or school, or missed a medical appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Worobey, PhD, DPT, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Information will be shared throughout duration of collaboration.
Access Criteria: A request will be made to the Principal Investigator, who will consider the request. No identifiable information will be shared.